CLINICAL TRIAL: NCT05749952
Title: Digital Weight Bearing Shape Capture Socket Technology to Preserve Limb Health and Improve Rehabilitation Outcomes
Brief Title: Digital Weight Bearing Shape Capture Socket Technology
Acronym: DWB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Sashwati Roy, Professor of Surgery, Indiana University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 15478
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Amputation; Prosthesis User; Residual Limbs

STUDY DESIGN:
Intervention Model Description: This is a crossover study where participants perform baseline visit in standard of care and then switched to DWB arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Symphonie Aqua System - Non-Digital (Socket B) (Experimental): A digital weight bearing test socket where shape capturing is done in full weight bearing
  Interventions: Device: Symphonie Aqua Digital System mediated sh
- Standard of Care (SoC) (Active Comparator): This is standard of care socket design where sockets are fabricated in non-weight bearing position
  Interventions: Device: Symphonie Aqua Digital System mediated sh

INTERVENTIONS:
Device: Symphonie Aqua Digital System mediated sh — For socket fabrication, the shape capturing is done in full weight bearing.

SUMMARY:
The study will determine if Symphonie Aqua Digital System, a new method of socket creation, in a weight-bearing environment, may produce more successful fitting and comfortability & functional outcomes than traditional sockets (non-weight bearing scanning). Additionally, the study will determine if a well-fitting socket will positively impact the overall health of amputee residual limb.

DETAILED DESCRIPTION:
This study will compare the use of Symphonie Aqua Digital System, which is a new way to create a socket for prosthetics, to the current method that is generally used to create sockets. The study will look at the differences in comfort and fit between the Symphonie Aqua Digital System and the current standard of care (SOC).

The study will determine if Symphonie Aqua Digital System, a new method of socket creation, in a weight-bearing environment, may produce more successful fitting and comfortability & functional outcomes than traditional sockets (non-weight bearing scanning). Additionally, the study will determine if a well-fitting socket will positively impact the overall health of amputee residual limb.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and above
* Unilateral trans-tibial amputees
* Ambulate at a K3 level or higher
* At least 3 months post-amputation per physician discretion
* Trans-tibial limb length greater than 4.5 inches in length
* Able to follow directions and independently give informed consent
* Must be able to ambulate without assistance

Exclusion Criteria:

* Age < 18 years
* Conditions that prevent wearing a prosthetic socket
* Soc Socket made with weight bearing system
* Cognitive deficits or mental health problems that would limit ability to consent and participate fully in the study protocol
* Women who are pregnant or who plan to become pregnant in the near future
* Weight > 280 lbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sashwati Roy, PhD., Principal Investigator — Indiana University
Locations (1):
- Indiana University Health Methodist Hospital, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SoC (Socket A) First, Then Symphonie Aqua System - Non-Digital (Socket B): Symphonie Aqua Digital System: A non-digital weight-bearing socket be used to create the check socket (temporary socket), which will be used to create a laminated final socket for home use and research outcomes. The check socket is temporarily used; whereas, the final socket is for long-term use.
  Soc Socket is a standard of care socket fabricated under non weight nearing position.
  The two groups are combined because all subjects started with SoC and then crossed over to Socket B.
Period: Standard of Care Socket
Arm/Group | SoC (Socket A) First, Then Symphonie Aqua System - Non-Digital (Socket B)
Started | 10
Completed | 10
Not Completed | 0
Period: Symphonie Aqua System - Non-Digital
Arm/Group | SoC (Socket A) First, Then Symphonie Aqua System - Non-Digital (Socket B)
Started | 10
Completed | 8
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: This is a longitudinal study where all participants first participated in standard of care arm and later on crossed over to test arm
Groups:
- Symphonie Aqua System - Non-Digital (Socket B): Socket shape capturing done under full weight bearing conditions, this is the test socket.
Arm/Group | Symphonie Aqua System - Non-Digital (Socket B)
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Trans-Epidermal Water Loss (TEWL)
Description: Differences between two systems and effects on Trans-Epidermal Water Loss (TEWL) will be measured by placing a non-invasive probe on the surface of the skin. Each measurement takes approximately 7-30 seconds each. The data is presented as g x m^-2xh^-1. Higher number indicates worse outcome.
Time Frame: 6 weeks
Population: Good quality TEWL data was available from n=5 in SoC and n=3 in DWB participants
Measure: Mean (Standard Deviation); unit: g x m^-2xh^-1
Groups:
- Socket A - Standard of Care Socket: SoC Socket is a standard of care socket fabricated under non-weight-bearing position.
- Socket B - Symphonie Aqua Digital System: Symphonie Aqua Digital System: A non-digital weight-bearing socket will be used to create the check socket (temporary socket), which will be used to create a laminated final socket for home use and research outcomes. The check socket will be temporarily used, whereas the final socket is for long-term use.
Arm/Group | Socket A - Standard of Care Socket | Socket B - Symphonie Aqua Digital System
Number analyzed (Participants) | 5 | 3
g x m^-2xh^-1 | 22.9 (9.46) | 14.7 (5.11)

2. Secondary Outcome: Laser Speckle Imaging (LSI)
Description: Differences between two systems and effects on blood flow will be measured using Laser Speckle Imaging (LSI) which is a non-invasive machine that uses light to capture the blood flow of participants residual limb. The blood flow (perfusion) data is expressed as perfusion units (PU) where PU is a relative, dimensionless measure of tissue blood flow or microvascular perfusion. Higher value indicates better perfusion (increase in blood flow).
Time Frame: 6-weeks
Measure: Mean (Standard Deviation); unit: PU
Arm/Group | Socket A - Standard of Care Socket | Socket B - Symphonie Aqua Digital System
Number analyzed (Participants) | 7 | 7
PU | 4.8 (3.4) | 4.1 (2.8)

3. Secondary Outcome: In-socket Pressure
Description: Measurements of socket pressure will be evaluated using in-socket sensors, which are positioned into the socket and function to detect the amount of residual load (pressure) that is placed on the limb.
Time Frame: 6-weeks
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Socket A - Standard of Care Socket | Socket B - Symphonie Aqua Digital System
Number analyzed (Participants) | 8 | 8
kPa | 1.93 (1.36) | 0.91 (0.79)

4. Secondary Outcome: Mobility (6MWT)
Description: 6-minute walking test (6MWT); Subject will walk for 6 consecutive minutes and, once the 6 minutes has elapsed, the distance covered will be measured.
Time Frame: 6-weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Socket A - Standard of Care Socket | Socket B - Symphonie Aqua Digital System
Number analyzed (Participants) | 8 | 8
meters | 376 (57) | 364 (47)

5. Secondary Outcome: Balance During Ambulation (TUG)
Description: Timed up and go test; In the timed up-and-go outcome, the patient rises from a seated position, walks three meters at a self-selected speed, turns around, and returns to the chair where they reseat themselves.
Time Frame: 6-weeks
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Socket A - Standard of Care Socket | Socket B - Symphonie Aqua Digital System
Number analyzed (Participants) | 8 | 8
Seconds | 9.3 (2.3) | 9.6 (2.0)

ADVERSE EVENTS:
Time Frame: 12-weeks
Arm/Group | Socket A - Standard of Care Socket | Socket B - Symphonie Aqua Digital System
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT05749952/Prot_SAP_001.pdf
  • Informed Consent Form (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT05749952/ICF_000.pdf